CLINICAL TRIAL: NCT06676592
Title: Digitally Acquired 3D Framework With Superimposed Preoperative Imaging Data for Intraoperative Guidance
Brief Title: A Study of the Use of 3D Technology to Guide Head and Neck Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-191
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Surgery; Head and Neck Disorder
Keywords: head and neck surgery; Scaniverse app; Memorial Sloan Kettering Cancer Center; 24-191

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants scheduled for head and neck surgery (Experimental): Participants are scheduled to undergo head and neck surgery in the Surgery Head and Neck Service at MSK
  Interventions: Diagnostic Test: Preoperative imaging; Diagnostic Test: 3D framework

INTERVENTIONS:
Diagnostic Test: Preoperative imaging — Preoperative imaging will be performed as part of the standard of care. Imaging data from US, CT, MRI, and/or PET performed for routine care will be used for this study.
Diagnostic Test: 3D framework — 3D images of surface landmarks will be acquired by use of US and the Scaniverse app before surgery, in conjunction with the participant's standard-of-care US or US-guided biopsy procedure

SUMMARY:
The purpose of this study is to test how the new 3D technology can be used to help improve the surgeon's ability to use information from standard imaging scans to guide head and neck surgery. Researchers will use the Scaniverse app during a standard ultrasound to create 3D images of participants' head and neck before their standard surgery. Researchers will see if the creation of a 3D framework profile with superimposed standard imaging scan information can be useful to the surgeon for guiding head and neck surgery

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Scheduled to undergo head and neck surgery in the Surgery Head and Neck Service at MSK

  o Note: If, for some reason, the participant is not scheduled to have standard preoperative imaging procedures, then the participant will have an ultrasound of the head and neck for research purposes.
* Scheduled to undergo standard of care preoperative imaging (ie, ultrasound (US), computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET)) in the Radiology Service at MSK
* Ability to understand and sign (or their legally acceptable representative (LAR) must sign) the written informed consent

Exclusion Criteria:

* Previous head and neck surgery or head and neck radiation
* Any condition which, in the judgement of the clinical investigator or his designee, might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of standard of care imaging studies successfully superimposed into 3D study framework for all participants | 1 year
  The primary objective of this study is to develop the technology of a 3D framework profile with superimposed preoperative imaging for intraoperative use. The process of developing the imaging technique will be considered successful if the imaging techniques and the hardware used are able to superimpose information from standard of care imaging studies into the 3D study framework for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Patel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent form), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org